CLINICAL TRIAL: NCT00643331
Title: The Effect of Exercise in Postmenopausal Women with Low Bone Density
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Swisse Vitamins Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2001.075
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2008-03

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteoporosis; Exercise; Low bone density; Falls
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise performed at the gym and at home
  Interventions: Behavioral: Exercise
- 2 (No Intervention): Usual care no additional exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise performed at gym and at home comprising strength, balance and impact exercise
  Arms: 1

SUMMARY:
This clinical trial aims to evaluate the effects of a 12 month gym- and home-based exercise program on bone density and falls risk factors in postmenopausal women with low bone density. It is hypothesised that the exercise program will lead to improvements in bone density and falls risk factors such as balance and muscle strength compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Be aged greater than 50 years
* Be at least 5 years post menopause (defined as the last normal menstrual bleed)
* Have osteopenia of the hip defined as a DXA T-score between -1 and -2.5 in one or more regions of the proximal femur (total hip, neck or trochanter regions).
* Have primary osteopenia
* Be community dwelling (not in residential care)
* Be able to attend an exercise program 3 times per week over the 12-month period
* Be able to read and write English

Exclusion Criteria:

* Secondary causes of bone loss such as osteomalacia, glucocorticoid medication
* Co-morbidities that would interfere with participation in exercise such as severe heart or pulmonary disease, inflammatory joint disease, severe osteoarthritis, psychiatric condition
* Physical or orthopaedic disabilities that would place the subject at risk or limit their ability to perform exercise
* Spinal osteoporosis defined as DXA T-score <-2.5
* A past vertebral fracture
* Body mass index > 35 or < 18.
* Currently on hormone replacement therapy (HRT)
* Current smoker
* Past use of HRT within the past 3 years and for more than 6 months duration
* Taking medication known to affect bone including oestrogen or steroid hormones
* Known clinically significant liver or renal disease
* Cancer within the past 5 years
* Doing regular strength training and/or weight-bearing exercise at least once per week in past 6 months
* Unlikely to comply with the intervention protocol

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2001-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Bone density measured using DXA at the lumbar spine and proximal femur | 12 months

SECONDARY OUTCOMES:
Falls risk factors | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Bennell, PhD, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia